CLINICAL TRIAL: NCT04578145
Title: Randomized Community Trial Community Based Screening for HIV Self Testing in Female Sex Workers in 23 Priority Districts in Indonesia (CBS HIVST in FSW)
Brief Title: Community Based Screening for HIV Self Testing in FSW in 23 Priority Districts in Indonesia
Acronym: CBS-FSW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kerti Praja Foundation (Other)
Collaborators: United Nations (Other)
Responsible Party: Principal Investigator, dr. Pande Putu Januraga, DrPH, Principal Investigator, Kerti Praja Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IDN09MHH
Record Dates: First submitted 2020-09-13; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Assisted community screening; Community based screening (CBS); Community HIV screening; Female sex worker (FSW); HIV self-testing; Human immunodeficiency virus (HIV); Oral fluid test (OFT); Outreach; Peer leader (PL); Unassisted community screening
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Stratified randomization was carried out in 23 priority districts involved.
  Kind of HIV testing offered for FSW intervention group is difference with those, in control group. Both HIV blood test and self-testing are implemented in the intervention group while it is just HIV blood test provided for the control one. For assisted in the intervention group, FSW been reached is offered HIV blood test at least 3 times at stages of outreaching process, before answering the eligibility questions and before watching the guided OFT self-testing video. If she receives, she will be accompanied to take the test in health facilities. If she refuses, she will be offered to perform or continue to take OFT self-testing. For unassisted, FSW only has an option to undertake OFT self-testing. The FSW accesses the link on website (www.teman-kita.org) and registers herself independently without assistance of outreach workers (OW) who usually offer HIV blood test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Female sex workers (FSW) (Other): Female sex workers (FSWs) community is the only group which has implemented the study intervention. This group has been underlined as the one of key affected populations (KAPs) that hold an increasing number of HIV incidence and prevalence recently in Indonesia even though it is approximately 226,791 FSWs by 2016 and around 5,254,065 clients access their services per year (MoH, 2017). The condition will be worst because the transmission definitely will continue to clients' sexual partner and moreover, their babies if their HIV status has not been known earlier. It means that lowering the transmission of HIV infection for FSWs, it will simultaneously lower its transmission to their sexual partners and furthermore their babies.
  Interventions: Diagnostic Test: HIV self-testing among female sex workers

INTERVENTIONS:
Diagnostic Test: HIV self-testing among female sex workers — Barriers faced by FSWs in terms of undergoing HIV blood test seemingly overcome through the implementation of alternative strategy of testing, by using OFT self-testing (Ora-Quick).
  Ora-Quick test used in this study measures antibody in oral fluid of participants. The oral fluid is collected used a test swab from participant's gum by wiping upper and lower gums once. The specimen mixed with buffered developer solution in test tube. Test result will appear in a short time, by 20 to 40 minutes and leading to interpret.
  Other Names: Community screening intervention

SUMMARY:
Indonesia is not yet on course to end HIV and AIDS by 2030. Epidemic transmission of HIV infection among key affected populations (KAPs), specifically FSWs, crucially has contributed to not achieving the target. Although the number of HIV tests performed annually has grown steadily in recent years, reaching 3,077,653 in calendar year 2018, pregnant women is accounted for a fairly large proportion of an increased number of persons being tested (MoH, 2018).

Regarding the FSWs, it has been a significant challenge to increase HIV testing uptake among this population. The challenge has been affected by Indonesia's national policy to close brothels. As consequence, many FSWs have become hidden and hard to reach. The implementation national policy also impacts on the way of commercial sex transactions in which it becomes underground, especially many FSWs utilize the new popularity of digital platforms to sell sexual services. It needs more effective case finding strategies to be implemented to reach them accordingly.

If it is considered from the FSWs side, there are some barriers to access HIV test services according to several reports. They consist of lack of money, time, stigma, discrimination, low-risk perception, fear, lack of accessibility, reluctance of health service providers to offer HIV testing and limited human resources. Oral fluid HIVST using is an alternative to traditional HIV testing services in the facility or other healthcare provider testing (UNAIDS, 2016). For this study, OraQuick is used as an alternative strategy for HIV testing among FSWs.

The primary objectives of this study are to assess whether proportion of FSW, who know their HIV status, increases or not; whether introduction of Oral fluid test increases the number of HIV testing at health facilities or not; and whether "assisted" or "unassisted" community HIV screening have a result to an increasing proportion of HIV testing at health facilities or not. Furthermore, CBS study aims to assess whether "assisted" and "unassisted" community HIV screening results to an increasing number of HIV positive case finding or not; and whether community HIV screening increases proportion of initiation of antiretroviral therapy (ART) or not. The secondary objectives of this study, meanwhile, are to measure acceptability of community-based self-screening in participation and to measure satisfaction of FSWs, who has participated, towards the delivery of community-based self-screening.

Regarding the inclusion criteria of this study, participant must be women 18 years old or older at enrollment; has a transactional sex (vaginal, oral and/or anal) at least once in the past month; does not uptake HIV test in the last 6 months; and acknowledges her HIV status 'negative' or 'unknown'. There are several exclusion criteria, which are FSW does not able to fulfill one of inclusion criteria that has been explained above; FSW does not has desire to participate due to several reasons; and she is currently participating in another HIV prevention study.

Outcome variables of this study are to compare the characteristic FSWs who receive self-testing and blood testing; who receive assisted and unassisted self-testing. Moreover, it compares the proportion of taking confirmatory test out of those who receive the test in the assisted and unassisted self-testing; proportion of FSWs who receive HIV test out of those who got offered for the test (including self-testing) in the intervention group with proportion of FSWs who receive HIV test in the control group; the proportion of FSWs taking confirmatory test (including self-testing) out of those receive the test in intervention groups and control group. It compares, furthermore, the proportion of HIV positive in the assisted, unassisted (intervention) and HIV positive in the control group. This study also compares ART initiation in the assisted, unassisted (intervention) and the control group. Additionally, it compares stigma scores and FSWs who went to a health facility for HIV testing between assisted, unassisted group and compares the HIV and STI risk behaviors between assisted and unassisted group. It calculates, lastly, the cascade of HIV testing and treatment.

DETAILED DESCRIPTION:
A. Background

1. The HIV Epidemic in Indonesia

   Until recently, Indonesia was among the few countries in which annual numbers of new HIV infections continued to rise (MoH, 2016). The latest epidemic modeling update indicated that except among men who have sex with man (MSM), annual numbers of new HIV infections had stabilized and begun to decline. However, with the current epidemic trajectory there would still be over 40,000 new HIV infections in the year 2030 (MoH,2016). Therefore, Indonesia is not yet on course to end HIV and AIDS by 2030.

   Although there has been a significant increase in the number of persons being treated for HIV/AIDS, the 108,479 people receiving ART as of December 2018 amounts to only 17 percent of the estimated number of people live with HIV (PLHIV) in the country (MoH, 2018). This makes Indonesia a performance "outlier" when compared to countries at comparable levels of gross national income (GNI) and health system development. The lack of more rapid progress has recently led key development partners to question Government of Indonesia (GOI) commitment to meaningfully addressing HIV and AIDS.

   Insufficient HIV testing remains a barrier to increasing ART coverage. The number of HIV tests performed annually has risen steadily in recent years, reaching 3,077,653 in calendar year 2018 (MoH, 2018). However, pregnant women account for a sizeable proportion of the increased number of persons being tested. While commendable, the case detection "yield" from testing pregnant women is relatively low. More effective case finding strategies need to be implemented to reach population sub-groups with higher HIV incidence and prevalence, including key affected populations (KAPs) such as female sex workers (FSW). Unless Indonesia can significantly increase its volume and efficiency of HIV testing, it will not be able to reach the first "95" of the UNAIDS 95-95-95 framework - that is, 95% of PLHIV know their HIV status.

   The main rationale is Indonesia's concentrated epidemic transmission of HIV infection among KAPs, specifically FSWs. In 2016 it is estimated that there are 226,791 female sex workers and around 5,254,065 clients access their service per year (MoH, 2017). This mode of transmission continues to clients' sexual partner and moreover, their babies. Lowering the transmission of HIV infection from FSW to their clients would simultaneously lower its transmission to their sexual partners and furthermore their babies.

   FSW can be grouped by "direct" (i.e., brothel-based) and "indirect" status with regard to way of selling their sex services. In 2016, however, the estimated number of FSW was not grouped into direct and indirect because it was considered that most of FSWs had shifted to becoming indirect due to Indonesia's national policy to close brothels. Due to this policy, most FSWs have become hidden and hard to reach, thus increasing the challenge of increasing HIV testing uptake among this sub-population. Many commercial sex transactions have become underground, especially given the new popularity of digital platforms to sell sexual services. This phenomenon has created a new demand to identify alternative strategies for increasing HIV testing uptake among FSW.
2. HIV Testing Among FSW

   Community based HIV-testing has been implemented in some countries such as Vietnam (Nguyen et al., 2019), Uganda (Ortblad et al., 2018), Malawi and Zimbabwe (Napierala et al., 2019). Non-governmental organizations in Indonesia had conducted study or pilot project on HIV test in men who have sex with men (MSM) outside health facility (Hidayat et al., 2019). This study was done to find an alternative to facility-based HIV testing, however MoH has been rather conservative in supporting non-health facility-based approach outside of mobile clinic testing which involves trained healthcare professional to perform HIV testing procedure according to the algorithm developed by the government. Mobile clinic testing strategy gave out insufficient result, especially in terms of linking those with positive HIV result for further follow-up and initiation of treatment. Cost-effectiveness of this approach was also doubted, at least in Jakarta (Cantelmo et al., 2019). This study found that the cost needed for mobile testing to identify at least one HIV positive case among FSW was almost six-times fold higher compared to finding similar target among transgender and MSM, and seventeen-times fold higher than those for identifying one HIV positive case among people who inject drugs (PWID). For the effective use of resource, this study suggested modification of the test frequency, time, and location for FSWs in Jakarta. In addition, this study also recommended the need for alternative strategies to increase HIV test uptake among FSW.

   FSWs community are at greater risk of not only HIV infection, but also stigma, discrimination and violence. They first face stigma and discrimination due to engaging in sex work itself, or from HIV stigma, particularly in contexts of HIV burden, which later affect their access to HIV testing (UNAIDS, 2016). The latest World Health Organization (WHO) guidelines have highlighted HIV self-testing (HIVST) as important tool to identify more people with undiagnosed HIV and at high risk of HIV infection. Protection of privacy and confidentiality is one of the advantages of this modality which allows for removing stigma as barriers to access services. HIVST has been shown to be acceptable across varieties of population globally including for FSWs community (King et al, 2013). Oral fluid HIVST is an alternative to traditional HIV testing services in the facility or other healthcare provider testing (UNAIDS, 2016).
3. Role of Outreach Worker in HIV Self-testing Using Assisted and Unassisted Method

   In a study which assessed implementation and scale-up to HIV self-testing programs for female sex workers in Malawi and Zimbabwe, there were difference in preferences for how to access HIV self-testing, depended on how supportive the existing program infrastructure was (Napierala et al., 2019) In Zimbabwe, where there was a detailed understanding of the context of female sex workers and a ready framework to implement and evaluate HIV self-testing strategies, high acceptability (76%) and high accuracy of HIV self-testing was reported (Napierala et al., 2019). In contrast, peer-distribution models were favored by female sex workers in Malawi and female sex workers in Zimbabwe who were not engaged in the program (Napierala et al., 2019). Another study in Kampala (Uganda) evaluated HIV self-testing performance and results interpretation among FSWs who performed unassisted HIV self-testing, showed that misinterpretation of HIV self-test results were common among FSWs: 23% (12/56) of FSWs interpreted HIV-negative self-test results as HIV positive and 8% (3/37) of FSWs interpreted HIV-positive self-test results as HIV negative (Ortblad et al., 2018). The concordance between FSWs' instructions was 73% (95%CI 56% to 86%) for HIV-positive self-tests and 68% (95%CI 54% to 80%) for HIV-negative self-tests (Ortblad et al., 2018). This finding suggested training on use and interpretation of HIV self-test for the unassisted method might be necessary to prevent errors and to avoid the negative consequences of false-positive and false-negative HIV self-test results among FSWs.
4. Study Purpose

The study proposed in this protocol directly addresses the need to get more Indonesian FSW to "know their status" by providing an alternative, convenient HIV testing option in non-threatening community settings. In the Indonesian context where a reactive HIV test result using the MoH-mandated triple rapid test algorithm is needed to qualify for GoI-financed ART, community screening is seen as a mechanism for enabling FSW to conveniently determine their status and a facilitation mechanism for taking action based upon the community screening result, whether that entail going to a health facility for a confirmatory test in the case of a reactive screening result or adopting stronger prevention measures in the case of a non-reactive screening result, including Pre-Exposure Prophylactic (PrEP) as this prevention method is rolled out in Indonesia.

The study will produce scientifically strong evidence as to whether two alternative models of community HIV screening among FSW (assisted and unassisted) result in (1) increased rates of formal HIV testing at health facilities and (2) increased rates of treatment initiation in districts in which the community screening intervention is added to the existing FSW community outreach model.

Two alternative study protocols are described in this document. The bulk of this document presents a protocol for a community randomized controlled trial (cRCT), which is the preferred research design option. However, due to a delay in procurement of the OraQuick® rapid HIV test kits that are to be used in the study, there may be insufficient time to undertake a full cRCT. Accordingly, a contingency protocol that can be implemented in a shorter period of time is also presented.

B. Study Design

1. Design Summary

   The study will be undertaken in the 23 "acceleration" districts in the National AIDs Program. These are: Kota Medan, Deli Serdang, Kota Palembang, Kota Bandar Lampung, Kota Tangerang Selatan, Tangerang, Kota Jakarta Selatan, Kota Jakarta Timur, Kota Jakarta Pusat, Kota Jakarta Barat, Kota Jakarta Utara, Bogor, Kota Bekasi, Kota Bandung, Kota Depok, Kota Semarang, Kota Surakarta, Kota Malang, Kota Surabaya, Kota Denpasar, Kota Makassar, Kota Sorong and Kota Jayapura. These are districts with high HIV prevalence among HIV key populations, including FSW, and have comprehensive ongoing HIV-TB intervention packages consisting of both health services and community prevention and support programs. As for the FSWs program, these 23 priority districts already implementing a comprehensive outreach package (reach to test and simplified case management for FSWs living with HIV).
2. Randomization

   Stratified randomization was carried out for the 23 priority districts involved in this study. First, sampling strata were created by sorting the mean average value of achieved HIV testing target per semester from 2018-2019 in each district from the largest to the smallest. The second step was to sort the districts into eight groups of three districts, except for the last group which will only consist of two districts. Randomization for intervention and comparison group were then carried out within these groups of eight with 2:1 ratio (2 intervention: 1 comparison).
3. Recruitment and Sample Size

All FSW in intervention districts who meet study eligibility criteria will be offered community screening. FSW in comparison districts will continue to receive the current standard package of interventions.

In to be able to detect a 10 percentage point difference in the rate of HIV testing at health facilities between FSW in intervention vs. comparison districts and have 95% certainty that a difference of that magnitude would not have occurred by chance and 90% certainty of detecting a difference of this magnitude if the difference was real/"the truth," the following sample of FSW will be needed in intervention and in comparison districts:

n ≥ [Z1-α (2P(1-P))1/2 + Z1-β (P1(1-P1) + P2(1-P2)2 / (P1-P2)2] * deft

Where:

Z1-α = the Z score for the level of statistical confidence, or statistical precision, desired (for 95%, Z = 1.96) Z1-β = the Z score for the desired statistical power (for 90% one-sided test, Z = 1.282) P1 = the expected population proportion in the comparison group of districts (set = 0.5 - this is the worst-case scenario and will produced a sample size that is adequate irrespective of the actual proportion P2 = the expected population proportion in the intervention group of districts (set = 0.6 - assume minimum effect size to be realized of 10 percentages points) P = (P1-P2) / 2 (P1-P2) = the magnitude of comparison-group differences (or change over time) to be detected with the specified level of precision and power (assumed to be +/- 10 percentage points) deft = design effect to compensate for clustering at the district level (1.5 assumed).

The required sample size is thus n ≥ 635 per experimental group; ≥ 761 after 20% allowance for lost-to-follow up Interpretation: we would need to recruit 761 FSW who self-test for HIV testing in the intervention districts and 761 FSW for HIV testing at health facilities in comparison districts to be able to detect a 10 percentage point difference in the rate of HIV testing at health facilities (intervention vs. comparison districts) to have 95% certainty that a difference of that magnitude would not have occurred by chance and 90% certainty of detecting a difference of this magnitude if such a difference existed.

In order to assess whether "assisted" or "unassisted" community HIV screening among FSW results in a larger increase in the rate of HIV testing at health facilities, we would need samples of size n ≥ 761 each of FSW who received assisted and unassisted screening in intervention districts, a total of n ≥ 1,522 FSW in intervention districts, plus n ≥ 761 in comparison districts.

Sample size requirements for the third question measurement pertains to the number of FSW who test positive for HIV at a health facility and are thus eligible to initiate treatment. This will depend upon (1) the number of FSW presenting at health facilities for testing and (2) the positivity rate among those tested. Sample sizes should thus be calculated accordingly. If we assume a testing positivity rate of 3%, it is apparent that the expected number of FSWs who would be eligible for treatment will be small and we will lack sufficient statistical power to make meaningful comparisons with comparison districts. For this reason, it is recommended that the impact of community screening among FSW be measured using system information HIV and AIDS data (SIHA) for FSW in both intervention and comparison districts. This estimate of impact derived in this way will be confounded if it were to be the case that interventions other than HIV self-testing were to be better implemented in intervention vs. comparison districts. It might be possible to minimize this potential bias by including measures of intervention implementation performance in the intervention and comparison districts in multivariable analyses. Thus, a large enough sample size is required to ensure sufficient power to determine the difference in the intervention and control districts.

C. The Intervention

1. General Description of The Intervention

The community screening intervention will be implemented as an additional component to be added in intervention districts to the intervention package currently being implemented by UNFPA's Implementation Units (IUs). In "control districts" implementation of the UNFPA-supported GFATM will proceed without modification as concerns community screening.

D. Data Collection Protocols

1. Baseline survey

   An application will be developed so that the survey can be completed and submitted to a server using mobile phones Outreach worker (OW)/Peer educator (PE)/Female sex worker (FSW). The following basic information will be gathered (see draft questionnaires for the baseline and post-test surveys in the annex of this protocol).
   * Name (full name/initial)
   * Age
   * Date of birth
   * Test Kit ID Number
   * Education
   * Marital status
   * Age at initiation of sex work
   * Number of clients last seven (7) days
   * Methods of clients' recruitment (fixed facility, street, internet, online platform)
   * Consistency of condom use
   * Ever been tested for HIV
   * When last time tested
   * Ever been diagnosed with an sexually transmitted infections/STI (other than HIV)
2. Post-test Survey

   The following inquiries will be made:
   * The clarity of information being provided (flier or short video), on a scale of 1-5
   * The easiness of test procedure, on a scale of 1-5
   * Perceived accuracy of the test result, on a scale of 1-5
   * The quality of response by the assigned contact person/hotline, on a scale of 1-5
   * Clients' acceptance/perception towards the study procedure
   * The likelihood of clients to recommend their peers to take the test, on a scale of 1-5
   * Test result
   * How likely is it that the client will get a HIV test at a health facility as a result of the community screening test, on a scale of 1-5
   * Comments and suggestions.
3. Routine Recording

Because of limitations in the data recorded and reported by health facilities, the study will rely primarily upon data recorded by IU outreach staff. Modifications will be made to the data recording and reporting systems currently being used to facilitate collection of the data needed for the study in a manner that minimizes additional recording and reporting burden. The nature of the adjustments to be made will be different for "assisted" and "unassisted" community screening.

For unassisted approach, additional information will be gathered as indicated below:

1. Numbers of FSW who access the link online
2. Numbers of FSW who are deemed eligible
3. Numbers of FSW who fill in baseline survey and agree to participate
4. Numbers of FSW who agree to take HIV test at health facility
5. Numbers of FSW who request the kit being delivered vs picking-up at fixed location
6. Numbers of FSW who upload the test result
7. Numbers of reactive vs non-reactive test result
8. Numbers of FSW who complete the post-test survey
9. Among FSW with community screening tests, the numbers that were subsequently tested at a health facility (reactive OR non-reactive)
10. Number of FSW initiating ART.

4. Numbering System for Test Kit and Other Instruments

1. Recording Test Kit ID

   Every test kit will have a unique ID number, which will later be referred to as the Kit ID number. The Kit ID Number is to be filled in on all instruments and forms that are to be linked to the test results (e.g., baseline survey, test results form, post-test survey, routine data record in each IU, etc.). This number needs to be identified at all times to make sure that each participant is only assigned to one test kit, matching the kit with the results, and to track the stock of the test kit remained. The format of this ID kit will be "01-001", where the first 2 digits are to identify the number of the district in which participants take the test, and the last 3 digits are to identify which test kit the participant is using. This test kit ID will also be later used for each IU to track the distribution of the test kit. Every test kit being distributed, either in a fixed place or delivered through same-day delivery services, will be recorded and tracked by each IU. An MS Excel or MS Access form will be developed to record and track the Kit ID Number.
2. Recording temporary FSW ID

   On the ground of confidentiality, participants' full name will not be revealed and used within this study. A new system to ensure the reliable yet confidential identification of study participants needs to be established. Every participant in the study will be assigned to a temporary FSW ID. The format will be the first 4 letters of participants' names added by the date of birth (yy/mm/dd). For example, a participant named "INDRIYANTI" who was born on March 5th, 1976, her temporary FSW ID will be "INDR760305". For FSW whose name contains only 3 letters, the number zero will be added after the last letter. For example, an FSW whose name is "AYU" and was born on March 5th1976, her temporary will be "AYU0760305". This temporary FSW ID will be used to ensure that each participant is only assigned to one test kit, to track test results, and to be filled in the baseline and post-test survey.
3. Matching Test Kit ID and temporary FSW ID

   To match the test kit ID and temporary FSW ID, an automatic system needs to be developed to detect it precisely. This way, we can be sure that each participant only gets to participate in this study once (from receiving the kit, performing the test, and reporting the result).
4. Paper Based Data Collection

In the event that participants' data are collected by paper, a procedure to upload the data into the established online system will be developed. Each data manager in the IUs needs to conduct the procedure regularly. This is to ensure that all data are being captured thoroughly.

E. Research Ethics and Permission

Participation in the study will be entirely voluntary. For the assisted testing, formal signed consent or witnessed verbal informed consent will be obtained by outreach workers. Records of informed consent will be managed /safeguarded using sealed envelope with unique number. To ensure the confidentiality, in the base line data only unique number will be recorded. A draft of the informed consent form can be found in Annex-3 of this protocol. For unassisted screening, every study participant should fill in the check box of website or application to provide consent: "By signing this form/ticking this box, I understand that I am thereby agreeing to enroll in this study" and test kit is not sent out if the check box is not checked by the user.

This protocol will be reviewed by the Faculty of Medicine Udayana University Institutional Review Board (IRB) prior to study initiation. Approval of the protocol in either its original or modified form is required.

Research permission will be submitted to Department of Internal Affairs Republic of Indonesia, which will subsequently be referred to the licensing office in each provinces and priority districts.

ELIGIBILITY:
Inclusion Criteria:

* Women, 18 years or older at enrollment
* Reports transactional sex (vaginal, oral and/or anal) at least once in the past month
* No HIV test in last 6 months
* Self-reported HIV negative OR HIV status unknown

Exclusion Criteria:

* Unwilling to participate for any reason
* Concurrently participating in another HIV prevention study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1522 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
HIV testing uptake | 7 months
  Number of FSWs receiving OFT and facility-based HIV testing, collected from OFT result (Annex 8) and blood test result (Annex 11).
HIV Positivity rate | 7 months
  Proportion of HIV positive cases among all FSWs who receive facility-based HIV testing (including those who receive post-OFT confirmatory testing), collected through blood test result form (Annex 11).
Antiretroviral (ARV) initiation rate | 7 months
  Proportion of FSWs with confirmed HIV positivity through facility-based testing (including post-OFT confirmatory tests) who initiate ARV treatment, collected through ARV initiation form (Annex 12).

SECONDARY OUTCOMES:
Age | at enrollment
  Continuous variable of participant's age, starting from 18, collected through baseline survey.
Education | at enrollment
  Categorical variable of educational level, collected from baseline survey.
Marital status | at enrollment
  Categorical variable of marital status, collected through baseline survey.
Client source | at enrollment
  Categorical variable of places where clients are obtained, collected through baseline survey.
Age of first sexual transaction | at enrollment
  Continues variable of participant's age, starts from 18, collected through baseline survey.
Condom use | at enrollment
  Frequency of condom use within the past month, collected through baseline survey.
Number of clients in the past 7 days | at enrollment
  Number of clients in the last 7 days, collected through baseline survey.
Primary partner | at enrollment
  Binary variable of reported primary partner in the past month, collected through the baseline survey.
History of HIV test | at enrollment
  Length of time since last HIV test, collected through baseline survey.
History of discomfort during sex or around genitalia within the past six months | at enrollment
  Reported history of discomfort during sex and/or around genitalia within the past six months (yes, no, unsure), collected through baseline survey.
History of sexually transmissible infections (ever been diagnosed with STI by a doctor within the past six months) | at enrollment
  History of having ever been diagnosed with STI by a doctor within the past six months (yes, no, unsure), collected through baseline survey.
Previous knowledge of OFT | at enrollment
  Categorical variable previous knowledge on OFT, collected through baseline survey.
Stigma score | at enrollment
  Likert scale of 1-5, 1 being strongly disagree and 5 being strongly agree, to statements in the 12-item short version HIV stigma scale by Reinius et al, 2017. Collected through baseline survey.
Clarity of OFT instructions | immediately after OFT, self-testing
  Likert scale of 1-5, 1 being very unclear and 5 being very clear, collected through post-test survey.
Peer or OW assistance during OFT | immediately after OFT, self-testing
  Binary variable of whether or not the FSW receives assistance from a peer/OW during OFT, collected through post-test survey.
Difficulty of OFT use | immediately after OFT, self-testing
  Likert scale of 1-5, 1 being very difficult and 5 being very easy, collected through post-test survey.
Difficulty of interpreting OFT results | immediately after OFT, self-testing
  Likert scale of 1-5, 1 being very difficult and 5 being very easy, collected through post-test survey.
Perceived support (only for assisted OFT) | immediately after OFT, self-testing
  Likert scale of 1-5, 1 being very unsupportive and 5 being very supportive, collected through post-test survey.
Willingness to receive routine testing after OFT (only for negative OFT) | immediately after OFT, self-testing
  Likert scale of 1-5, 1 being very unwilling and 5 being very willing, collected through post-test survey.
Experience of testing | immediately after OFT, self-testing
  Likert scale of 1-5, 1 being very unpleasant and 5 being very pleasant, collected through post-test survey.
Certainty of result | immediately after OFT, self-testing
  Likert scale of 1-5, 1 being very uncertain and 5 being very certain, collected through post-test survey.
OFT result | immediately after OFT, self-testing
  Categorical variables of OFT results (reactive, non-reactive and indeterminate), collected through post-test survey.
Desire to confirm OFT result | immediately after OFT, self-testing
  Likert scale of 1-5, 1 being very unwilling and 5 being very willing, collected through post-test survey.
Desire to recommend OFT testing to peers | immediately after OFT, self-testing
  Likert scale of 1-5, 1 being very unwilling and 5 being very willing, collected through post-test survey.

CONTACTS AND LOCATIONS:
Overall Officials: Anak Agung Sagung Sawitri, DR, Principal Investigator — Kerti Praja Foundation; I G. A. A Mahendra, MPH, Study Chair — Kerti Praja Foundation
Locations (1):
- Kerti Praja Foundation, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No
There is no sharing individual participant data (IPD) because researchers absolutely have an intention to protect their individual privacy. FSWs have also been explained that their data will not be shared for anyone. It has been emphasized clearly in inform consent.
  Moreover, concerning the stigmatization for FSWs who infected HIV across Indonesia, researches obviously restrict an access publicly for IPD. This is essential to increase self-esteem of FSWs in order to undergo HIV testing periodically.

REFERENCES:
- [Background] King EJ, Maman S, Bowling JM, Moracco KE, Dudina V. The influence of stigma and discrimination on female sex workers' access to HIV services in St. Petersburg, Russia. AIDS Behav. 2013 Oct;17(8):2597-603. doi: 10.1007/s10461-013-0447-7. PMID 23525789
- [Background] Napierala S, Desmond NA, Kumwenda MK, Tumushime M, Sibanda EL, Indravudh P, Hatzold K, Johnson CC, Baggaley RC, Corbett L, Cowan FM. HIV self-testing services for female sex workers, Malawi and Zimbabwe. Bull World Health Organ. 2019 Nov 1;97(11):764-776. doi: 10.2471/BLT.18.223560. Epub 2019 Sep 3. PMID 31673192
- [Background] Nguyen VTT, Phan HT, Kato M, Nguyen QT, Le Ai KA, Vo SH, Thanh DC, Baggaley RC, Johnson CC. Community-led HIV testing services including HIV self-testing and assisted partner notification services in Vietnam: lessons from a pilot study in a concentrated epidemic setting. J Int AIDS Soc. 2019 Jul;22 Suppl 3(Suppl Suppl 3):e25301. doi: 10.1002/jia2.25301. PMID 31321903
- [Background] Ortblad KF, Kibuuka Musoke D, Ngabirano T, Nakitende A, Taasi G, Barresi LG, Barnighausen T, Oldenburg CE. HIV self-test performance among female sex workers in Kampala, Uganda: a cross-sectional study. BMJ Open. 2018 Nov 8;8(11):e022652. doi: 10.1136/bmjopen-2018-022652. PMID 30413504
- [Background] Shahmanesh M, Patel V, Mabey D, Cowan F. Effectiveness of interventions for the prevention of HIV and other sexually transmitted infections in female sex workers in resource poor setting: a systematic review. Trop Med Int Health. 2008 May;13(5):659-79. doi: 10.1111/j.1365-3156.2008.02040.x. Epub 2008 Feb 11. PMID 18266784
- [Background] Shokoohi M, Karamouzian M, Khajekazemi R, Osooli M, Sharifi H, Haghdoost AA, Kamali K, Mirzazadeh A. Correlates of HIV Testing among Female Sex Workers in Iran: Findings of a National Bio-Behavioural Surveillance Survey. PLoS One. 2016 Jan 25;11(1):e0147587. doi: 10.1371/journal.pone.0147587. eCollection 2016. PMID 26807584
- [Background] Johnston LG, Bonilla L, Caballero T, Rodriguez M, Dolores Y, de la Rosa MA, Malla A, Burnett J, Terrero V, Martinez S, Morgan O. Associations of HIV Testing, Sexual Risk and Access to Prevention Among Female Sex Workers in the Dominican Republic. AIDS Behav. 2017 Aug;21(8):2362-2371. doi: 10.1007/s10461-016-1616-2. PMID 27896553
- [Background] Suthar AB, Ford N, Bachanas PJ, Wong VJ, Rajan JS, Saltzman AK, Ajose O, Fakoya AO, Granich RM, Negussie EK, Baggaley RC. Towards universal voluntary HIV testing and counselling: a systematic review and meta-analysis of community-based approaches. PLoS Med. 2013 Aug;10(8):e1001496. doi: 10.1371/journal.pmed.1001496. Epub 2013 Aug 13. PMID 23966838
- [Background] Tokar A, Broerse JEW, Blanchard J, Roura M. HIV Testing and Counseling Among Female Sex Workers: A Systematic Literature Review. AIDS Behav. 2018 Aug;22(8):2435-2457. doi: 10.1007/s10461-018-2043-3. PMID 29464430
- [Background] Tun W, Vu L, Dirisu O, Sekoni A, Shoyemi E, Njab J, Ogunsola S, Adebajo S. Uptake of HIV self-testing and linkage to treatment among men who have sex with men (MSM) in Nigeria: A pilot programme using key opinion leaders to reach MSM. J Int AIDS Soc. 2018 Jul;21 Suppl 5(Suppl Suppl 5):e25124. doi: 10.1002/jia2.25124. PMID 30033680
- [Background] Wariki WM, Ota E, Mori R, Koyanagi A, Hori N, Shibuya K. Behavioral interventions to reduce the transmission of HIV infection among sex workers and their clients in low- and middle-income countries. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD005272. doi: 10.1002/14651858.CD005272.pub3. PMID 22336811
- [Background] Reinius M, Wettergren L, Wiklander M, Svedhem V, Ekstrom AM, Eriksson LE. Development of a 12-item short version of the HIV stigma scale. Health Qual Life Outcomes. 2017 May 30;15(1):115. doi: 10.1186/s12955-017-0691-z. PMID 28558805
- [Result] Wirtz AL, Pretorius C, Beyrer C, Baral S, Decker MR, Sherman SG, Sweat M, Poteat T, Butler J, Oelrichs R, Semini I, Kerrigan D. Epidemic impacts of a community empowerment intervention for HIV prevention among female sex workers in generalized and concentrated epidemics. PLoS One. 2014 Feb 6;9(2):e88047. doi: 10.1371/journal.pone.0088047. eCollection 2014. PMID 24516580
- [Result] Batona G, Gagnon MP, Simonyan DA, Guedou FA, Alary M. Understanding the intention to undergo regular HIV testing among female sex workers in Benin: a key issue for entry into HIV care. J Acquir Immune Defic Syndr. 2015 Mar 1;68 Suppl 2:S206-12. doi: 10.1097/QAI.0000000000000452. PMID 25723986
- [Result] Bengtson AM, L'Engle K, Mwarogo P, King'ola N. Levels of alcohol use and history of HIV testing among female sex workers in Mombasa, Kenya. AIDS Care. 2014;26(12):1619-24. doi: 10.1080/09540121.2014.938013. Epub 2014 Jul 21. PMID 25040114
- [Result] Deering KN, Montaner JS, Chettiar J, Jia J, Ogilvie G, Buchner C, Feng C, Strathdee SA, Shannon K. Successes and gaps in uptake of regular, voluntary HIV testing for hidden street- and off-street sex workers in Vancouver, Canada. AIDS Care. 2015;27(4):499-506. doi: 10.1080/09540121.2014.978730. Epub 2014 Nov 27. PMID 25428563
- [Result] Dugas M, Bedard E, Batona G, Kpatchavi AC, Guedou FA, Dube E, Alary M. Outreach strategies for the promotion of HIV testing and care: closing the gap between health services and female sex workers in Benin. J Acquir Immune Defic Syndr. 2015 Mar 1;68 Suppl 2:S198-205. doi: 10.1097/QAI.0000000000000463. PMID 25723985
- [Result] Hidayat R, Marguari D, Hairunisa N, Suparno H, Magnani R. Community HIV Screening Among MSM in Three Indonesian Cities. Curr HIV Res. 2019;17(1):65-71. doi: 10.2174/1570162X17666190321115419. PMID 30907323
- [Result] Kerrigan DL, Fonner VA, Stromdahl S, Kennedy CE. Community empowerment among female sex workers is an effective HIV prevention intervention: a systematic review of the peer-reviewed evidence from low- and middle-income countries. AIDS Behav. 2013 Jul;17(6):1926-40. doi: 10.1007/s10461-013-0458-4. PMID 23539185
- [Derived] Yunus JO, Sawitri AAS, Wirawan DN, Mahendra IGAA, Susanti D, Utami Ds NKAD, Asanab D, Narayani IA, Mukuan OS, Widihastuti A, Magnani R, Januraga PP. Web-Based Multifaceted Approach for Community-Based HIV Self-Testing Among Female Sex Workers in Indonesia: Protocol for a Randomized Community Trial. JMIR Res Protoc. 2021 Jul 21;10(7):e27168. doi: 10.2196/27168. PMID 34287217
- See also: Indonesia Factsheet, UNAIDS - 2016 — http://www.unaids.org/sites/default/files/media_asset/UNAIDS_FactSheet_en.pdf
- See also: Karawita D.A. , Tennakoon S.U.B. , Suranga S. , Dissanayake M.S.W. Acceptability of Oral-fluid rapid HIV 1 and 2 antibody tes among selected key populations in Sri Lanka. Sri Lanka Journal of Sexual Health and HIV Medicine Volume 3. — http://doi.org/10.4038/joshhm.v3i0.59
- See also: World Health Organization, Consolidated guidelines on HIV testing services. 2015. Geneva, Switzerland: WHO. — https://apps.who.int/iris/bitstream/handle/10665/179870/9787564176464-chi.pdf

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT04578145/Prot_SAP_ICF_000.pdf